CLINICAL TRIAL: NCT04967144
Title: Right/Left Judgement in Carpal Tunnel Syndrome
Brief Title: Carpal Tunnel Syndrome, Right/Left Judgement
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeniz Akçay, Study Director, Bozyaka Training and Research Hospital
Other Study IDs: 2021/40
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome, body schema
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carpal Tunnel syndrome: .Patients with carpal tunnel syndrome
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Montreal Cognitive Assessment Test
- Control subjects: Healthy subjects
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Montreal Cognitive Assessment Test

INTERVENTIONS:
Diagnostic Test: Nerve conduction study — Participants with carpal tunnel syndrome will consist of individuals whose diagnosis has been confirmed by an electrophysiological study.
  Participants in the control group will consist of those who have been confirmed not to have carpal tunnel syndrome by nerve conduction study.
Diagnostic Test: Montreal Cognitive Assessment Test — Montreal Cognitive Assessment Test evaluates eight separate cognitive functions. Thirty is the highest score. The scores equal to or above 26 are considered normal cognitive function.

SUMMARY:
The discrimination of the right/left side of the body is related to the integrity of the motor and somatosensory areas at the cortical and subcortical levels. Although some studies have shown that there may be an effect on the right/left representation at the cortical and subcortical levels in cases that cause severe neuropathy and neuropathic pain, this effect has not been proven in milder neuropathies. In this study, the effect on right/left side discrimination will be investigated even in cases with carpal tunnel syndrome. Additionally, the investigators aimed to assess the relationship between right/left discrimination and symptom severity.

DETAILED DESCRIPTION:
The left/right discrimination is a motor imagery task that involves viewing images of a body part and determining whether each image belongs to the left or right side of the body or if it rotates towards it. Some studies have shown that there may be an effect on the right/left representation at the cortical and subcortical levels in cases that cause severe neuropathy and neuropathic pain, this effect has not been proven in milder neuropathies, such as carpal tunnel syndrome. In this study, the relationship between right/left decision accuracy will be compared with control subjects. The investigators will assess the relationship between right/left judgment and symptom severity, two-point discrimination, and handgrip force.

The hypothesis of the study are:

1. The right/left discrimination accuracy is less than the control subjects.
2. Right/left discrimination is in relationship with symptom severity, two-point discrimination, and handgrip force.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a duration of symptoms associated with unilateral CTS of at least 3 months
* Participants with clinically and nerve conduction study confirmed carpal tunnel syndrome
* All participants will be right-hand dominance and diagnosed with carpal tunnel syndrome on the same side
* Participants with MOCA score minimum 26.

Exclusion Criteria:

* Severe visual impairment that may prevent performing the test
* Polyneuropathy
* Cervical spine surgery history
* Presence of abnormal cervical spine, shoulder, and elbow joint examination findings
* Patients with any history of surgery for the upper extremity
* Congenital/Developmental upper extremity malformations
* Central nervous system disease
* Antihistaminic, gabapentinoids, antiepileptics, methylphenidate, modafinil, neuroleptics use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Carpal Tunnel Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Left/right judgement Task | 3 months
  The Recognize tablet application will be used within the scope of the 'Graded Motor Imagery' set, in the series of publications created by www.noigroup.com right/left side judgement. The application will be performed on a single tablet screen. Within the scope of the application, right and left-hand pictures will be shown to the participants in varying positions and angles at 5-second intervals. The test consists of 50 pictures. At the end of the test, the accuracy rate and the average reaction time will be calculated separately for the right and left sides.

SECONDARY OUTCOMES:
Handgrip strength | 3 months
  The both handgrip strength of the participants will be evaluated with a JAMAR hand dynamometer.
Two-point discrimination test | 3 months
  The participants will use a 2-point disc-criminator with 2-point separation and the narrowest interval reported by the participant as two separate points with repetitive measurements from the distal volar region of both index fingers will be recorded.
Visual Analogue Scale | 3 months
  The patient will be asked to mark his/her severity of pain on a 10-cm horizontal line with number 0 one end representing 'no' and number 10 on the other end indicating 'very severe pain'.
PainDETECT questionnaire | 3 months
  The presence of neuropathic pain will be evaluated with the painDETECT questionnaire. The maximum score is 35 and a high score indicates the severity of neuropathic pain. When the painDETECT questionnaire score is more than 13, it is indicated the presence of a neuropathic pain component.
Boston Carpal Tunnel Questionnaire | 3 months
  The questionnaire comprises two parts, the Symptom Severity (SSS) and the Functional Status Scale (FSS). In the SSS, there are 11 questions; responses may be scored one (mildest) point to five (most severe) points. In the FSS, there are eight questions assessing the difficulty in performing selected activities.

CONTACTS AND LOCATIONS:
Overall Officials: Seniz Akcay, Assoc Prof, Study Director — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Altinay Goksel Karatepe, Prof, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Fikriye Elif Saka, MD, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Asli Koskderelioglu, Assoc Prof, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Neslihan Eskut, Specialist, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital
Locations (1):
- University of Health Sciences Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The clinical study report will be shared at the end of the study.

REFERENCES:
- [Background] Breckenridge JD, Ginn KA, Wallwork SB, McAuley JH. Do People With Chronic Musculoskeletal Pain Have Impaired Motor Imagery? A Meta-analytical Systematic Review of the Left/Right Judgment Task. J Pain. 2019 Feb;20(2):119-132. doi: 10.1016/j.jpain.2018.07.004. Epub 2018 Aug 9. PMID 30098404
- [Result] Schmid AB, Coppieters MW. Left/right judgment of body parts is selectively impaired in patients with unilateral carpal tunnel syndrome. Clin J Pain. 2012 Sep;28(7):615-22. doi: 10.1097/AJP.0b013e31823e16b9. PMID 22688599
- [Result] Moseley GL. Why do people with complex regional pain syndrome take longer to recognize their affected hand? Neurology. 2004 Jun 22;62(12):2182-6. doi: 10.1212/01.wnl.0000130156.05828.43. PMID 15210879
- [Result] Williams LJ, Braithwaite FA, Leake HB, McDonnell MN, Peto DK, Lorimer Moseley G, Hillier SL. Reliability and validity of a mobile tablet for assessing left/right judgements. Musculoskelet Sci Pract. 2019 Apr;40:45-52. doi: 10.1016/j.msksp.2019.01.010. Epub 2019 Jan 24. PMID 30703633
- [Derived] Akcay S, Koskderelioglu A, Ince B, Elif Saka F, Eskut N, Goksel Karatepe A. Is the left/right judgment task performance altered in unilateral carpal tunnel syndrome: And associated with symptom severity? Musculoskelet Sci Pract. 2022 Dec;62:102641. doi: 10.1016/j.msksp.2022.102641. Epub 2022 Aug 4. PMID 35961062